CLINICAL TRIAL: NCT01851980
Title: Effects of Inhaled Furosemide on Breathlessness During Exercise in the Presence of External Thoracic Restriction: A Dose-Reponse Study
Brief Title: Inhaled Nebulized Furosemide & Physical Activity-Related Breathlessness
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: McGill University (Other)
Responsible Party: Principal Investigator, Dennis Jensen, Ph.D., Assistant Professor, McGill University
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 15-370-MUHC
Record Dates: First submitted 2013-05-07; First posted 2013-05-13 (Estimated); Last update posted 2017-02-14 (Actual); Status verified 2017-02

CONDITIONS: Breathlessness
Keywords: Furosemide; Exercise; Restrictive pulmonary disorder
MeSH Terms: conditions — Dyspnea; Motor Activity | interventions — Furosemide

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- CWS+Furosemide (40 mg) (Experimental): Chest wall strapping to reduce vital capacity by 20% of its baseline value + single-dose inhalation of furosemide (40 mg)
  Interventions: Other: CWS; Drug: Furosemide
- CWS+0.9% saline placebo (Placebo Comparator): Chest wall strapping to reduce vital capacity by 20% of its baseline value + single-dose inhalation of 0.9% saline placebo
  Interventions: Other: CWS; Drug: Placebo
- CWS+Furosemide (120 mg) (Experimental): Chest wall strapping to reduce vital capacity by 20% of its baseline value + single-dose inhalation of furosemide (120 mg)
  Interventions: Other: CWS; Drug: Furosemide

INTERVENTIONS:
Other: CWS — Chest wall strapping to reduced vital capacity by 20% of its baseline value
  Other Names: Chest wall strapping
Drug: Furosemide — 40 mg and 120 mg
  Arms: CWS+Furosemide (120 mg); CWS+Furosemide (40 mg)
Drug: Placebo — 0.9% saline
  Arms: CWS+0.9% saline placebo

SUMMARY:
Breathlessness on exertion is a common and troublesome complaint of individuals with restrictive lung disorders. In these adults, breathlessness contributes to physical activity-limitation and avoidance and an adverse health-related quality-of-life, often in a self-perpetuating cycle. It follows that alleviating dyspnea and improving exercise tolerance are among the principal goals in the management of adults with restrictive lung disorders. Nevertheless, effective management of breathlessness and physical activity-limitation remains an elusive goal for many healthcare providers and current therapies (e.g., antifibrotic agents, oxygen, exercise training) are only partially successful in this regard. Thus, research aimed at identifying breathlessness-specific medications to complement existing therapies for the management of physical activity-related breathlessness in restrictive lung disorders is timely and both clinically and physiologically relevant. The purpose of this randomized crossover study study is to examine the acute effects of two doses of inhaled nebulized furosemide (a loop diuretic) on the perception of breathlessness during laboratory-based cycle exercise in healthy, young men in the presence of an external thoracic restriction to mimic a 'mild' restrictive lung deficit. To this end, the investigators will compare the effects of inhaled 0.9% saline placebo and inhaled furosemide (40 mg and 120 mg) on detailed assessments of breathlessness (sensory intensity and affective responses) and its physiological determinants (ventilation, breathing pattern, dynamic operating lung volumes, cardio-metabolic function) symptom-limited, high-intensity, constant-work-rate cycle exercise testing with external thoracic restriction sufficient to mimic a 'mild' restrictive pulmonary deficit in healthy, men aged 18-40 years.

ELIGIBILITY:
Inclusion Criteria:

* Male
* Aged 18-40 years
* FEV1 ≥80% predicted
* FEV1/FVC >70%

Exclusion Criteria:

* Current or ex-smoker
* Body Mass Index <18.5 or >30 kg/m2
* Self-reported history of cardiovascular, vascular, respiratory, renal, liver, musculoskeletal, endocrine, neuromuscular and/or metabolic disease/dysfunction
* Taking doctor prescribed medications
* Allergy to sulfa medications

Ages: 18 Years to 40 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Estimated)
Dates: Start 2016-04; Primary Completion 2017-04 (Estimated); Study Completion 2017-09 (Estimated)

PRIMARY OUTCOMES:
Sensory intensity (Borg 0-10 scale) ratings of dyspnea at isotime | Participants will be followed until all study visits are completed, an expected average of 3 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Dennis Jensen, Ph.D., Principal Investigator — McGill University
Locations (1):
- Centre of Innovative Medicine of the McGill University Health Centre, Montreal, Quebec, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Clinical Exercise & Respiratory Physiology Laboratory (CERPL) of McGill University — http://www.mcgill.ca/cerpl